CLINICAL TRIAL: NCT04819256
Title: PACE-It Study : Primary Care Based Integrated Community Care Team Intervention to Improve the Health Outcomes of Patients Living With Diabetes and Complex Needs - a Feasibility Study
Brief Title: Primary Care Based Integrated Community Care Team Intervention
Acronym: PACE-It
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding diverted to expansion of programme and PACE-It App
Sponsor: SingHealth Polyclinics (Other)
Collaborators: Ministry of Health, Singapore (Other Government); Agency for Integrated Care, Singapore (Other); SingHealth Regional Health System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/2202
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Diabetes; Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes type2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Providers use PACE-It mobile application as a care co-ordination platform
  Interventions: Other: PACE-It mobile application
- Usual care (No Intervention): Providers use usual modes of communication (e.g., phone calls, emails)

INTERVENTIONS:
Other: PACE-It mobile application — Care co-ordination platform
  Arms: Intervention arm

SUMMARY:
PACE-It study is a non-blinded, mix-method randomized controlled trial within a single site. This study aims to test the feasibility of implementing a complex intervention comprising of a) a Primary Care Based integrated community care team delivery of person centered care, b) supported by a care co-ordination platform using a mobile application and its effectiveness in improving the glycemic control of patients living with Diabetes and have complex needs.

DETAILED DESCRIPTION:
PACE-It study aims to test the feasibility of implementing a complex intervention comprising of a) a Primary Care Based Community Care Team delivery of person centered care b) supported by a care co-ordination platform using a mobile application and its effectiveness in improving the glycemic control of patients living with Diabetes and complex needs.

This is a non-blinded, mix-method randomised controlled trial within the Marine Parade Community. The primary outcome will be glycemic control measure by the Glycated Haemoglobin (HbA1c). Secondary outcomes include blood pressure, LDL-cholesterol, Patient Activation Measure, Medication Adherence and Quality of Life. Data on patient and provider satisfaction and implementation process will be collected by the Qualitative method.

ELIGIBILITY:
Inclusion Criteria:

* Living within the designated geographical zone
* 50 years and above
* Satisfy the Medical Criteria below:

  1. Diabetes with HbA1c ≥ 9% (within past 6 months), and
  2. At least 1 complication

     1. chronic kidney impairment stage 3 and above, or diabetes overt nephropathy,
     2. ischaemic heart disease, or congestive cardiac failure,
     3. peripheral arterial disease, or diabetes foot/ diabetes foot-related complications,
     4. diabetic retinopathy/ treatment for retinopathy, and
     5. stroke, or transient ischaemic attack
* Satisfy at least 2 conditions in the psycho-social, functional or activation domain of which 1 criteria must be from the psycho-social domain:

  1. Psycho-social issues

     a. Lack of care giver support i. No care-giver (when indicated) ii. Care-giver skills gap/ stress iii. Inability of copy when patient is the care-giver b. Difficult relationships (family/ workplace/ social network) c. Social isolation/ lack of social connectivity i. Lives alone ii. Lack of social network support d. Financial i. Financial difficulty/ insecurity ii. Housing/ shelter issues iii. Poor money management
  2. Functional

     1. Clinical Frailty Score ≥ 4, requiring help in instrumental activities of daily living (iADL)
     2. Requires assistance in ADL or iADL
  3. Activation a. Lack of ability to manage health - disengaged or overwhelmed i. Anxiety or disease-related distress ii. Confusion or lack of understanding of care plans iii. Non-adherence to medications/ follow up
* Patient gives consent to participate
* For patients who may be seeing a Primary Care Physician (PCP) outside of the polyclinic for chronic disease management and where the PCP has indicated consent to co-manage the patient with the PACE-It team including the polyclinic physician
* Patient must be willing to receive care in the polyclinic

Exclusion Criteria:

* Patients who are on follow up with Primary Care Physicians or General Practitioners elsewhere for management of their chronic conditions and they do not consent to co-managing patient with the PACE-It team
* Patients who have severe cognitive impairment, depression or psychiatric conditions that interfere with the ability to engage with the healthcare team
* Patients who are (i) not community ambulant or (ii) bed bound
* Patients with terminal illness
* Patients who have are in other programs or research studies
* Patients who do not give consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | 1 year
  Glycemic control

SECONDARY OUTCOMES:
Blood pressure | 1 year
  Systolic and diastolic blood pressure (mmHg)
LDL-cholesterol | 1 year
  Low-density lipoprotein cholesterol
Patient activation measure (PAM) | 1 year
  Patient's activation levels
Medication adherence measure (MARS-5) | 1 year
  Patient's adherence to medication
EQ-5D-5L | 1 year
  Quality of life
Patient satisfaction | 1 year
  Qualitative survey and interview
Provider's satisfaction | 2 years
  Qualitative survey and interview
Cost-effectiveness | 2 years
  Cost-effectiveness of care model
Implementation of care model | 2 years
  Factors affecting implementation of care model

CONTACTS AND LOCATIONS:
Overall Officials: Sinead Zhen Wang, Dr, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics - Marine Parade, 80 Marine Parade Central, #01-792, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No